CLINICAL TRIAL: NCT02894931
Title: Effects of Dietary Interventions (Sugars, Amino Acids and Artificial Sweeteners) on Serum and Macrophage Atherogenicity
Brief Title: Effects of Dietary Interventions on Serum and Macrophage Atherogenicity
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Rambam Health Care Campus (Other)
Responsible Party: Principal Investigator, Prof. Tony hayek MD, Director, Department of Internal Medicine E, Rambam Health Care Campus
Allocation: Non-Randomized | Model: Crossover | Masking: None
Other Study IDs: 0285-16-RMB CTIL
Record Dates: First submitted 2016-08-22; First posted 2016-09-09 (Estimated); Last update posted 2016-09-27 (Estimated); Status verified 2016-09

CONDITIONS: Dietary Habits; Serum; Disease; Macrophage Atherogenicity; Atherosclerosis
Keywords: macrophage atherogenicity; dietary interventions; sugars; amino acids; artificial sweeteners; atherosclerosis
MeSH Terms: conditions — Feeding Behavior; Disease; Atherosclerosis | interventions — Monosaccharides; Disaccharides; Amino Acids; Sweetening Agents

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (15):
- Control (Sham Comparator): Dietary Interventions: Control- water, Flavered Chilled water, will be administered once after O.N fasting.
  Interventions: Other: Control- water
- Glucose (Active Comparator): Dietary Interventions: Glucose, Monosaccharides, at the dose of 50 g, based on oral loading tests, once.
  Interventions: Dietary Supplement: monosaccharides
- Fructose (Experimental): Dietary Interventions: Fructose, Monosaccharides, at the dose of 50 g, once.
  Interventions: Dietary Supplement: monosaccharides
- Galactose (Experimental): Dietary Interventions: Monosaccharides, at the dose of 50 g, once.
  Interventions: Dietary Supplement: monosaccharides
- Mannose (Experimental): Dietary Interventions: Monosaccharides, at the dose of 50 g, once.
  Interventions: Dietary Supplement: monosaccharides
- Maltose (Experimental): Dietary Interventions: The dose of the disaccharides - 50 g, once.
  Interventions: Dietary Supplement: Disaccharides
- Sucrose (Experimental): Dietary Interventions: The dose of the disaccharides - 50 g, once.
  Interventions: Dietary Supplement: Disaccharides
- Lactose (Experimental): Dietary Interventions: The dose of the disaccharides - 50 g, once.
  Interventions: Dietary Supplement: Disaccharides
- Saccharin (Experimental): Dietary Interventions: The dose of the different artificial sweeteners - 300 mg, is based on an average adult male body weight of 75 kg and is set not to exceed the acceptable daily intakes of saccharin, aspartame, sucralose and steviol that were reported at 15, 50, 5, and 4 mg/kg body weight/day by the USA Food and Drug Administration, once.
  Interventions: Dietary Supplement: Artificial Sweeteners
- Aspartame (Experimental): Dietary Interventions: The dose of the different artificial sweeteners - 300 mg, is based on an average adult male body weight of 75 kg and is set not to exceed the acceptable daily intakes of saccharin, aspartame, sucralose and steviol that were reported at 15, 50, 5, and 4 mg/kg body weight/day by the USA Food and Drug Administration, once.
  Interventions: Dietary Supplement: Artificial Sweeteners
- Sucralose (Experimental): Dietary Interventions: The dose of the different artificial sweeteners - 300 mg, is based on an average adult male body weight of 75 kg and is set not to exceed the acceptable daily intakes of saccharin, aspartame, sucralose and steviol that were reported at 15, 50, 5, and 4 mg/kg body weight/day by the USA Food and Drug Administration, once.
  Interventions: Dietary Supplement: Artificial Sweeteners
- Steviol (Experimental): Dietary Interventions: The dose of the different artificial sweeteners - 300 mg, is based on an average adult male body weight of 75 kg and is set not to exceed the acceptable daily intakes of saccharin, aspartame, sucralose and steviol that were reported at 15, 50, 5, and 4 mg/kg body weight/day by the USA Food and Drug Administration, once.
  Interventions: Dietary Supplement: Artificial Sweeteners
- Leucine (Experimental): Dietary Interventions: The dose of the different BCAAs Amino acids- 5 g, is set not to exceed the mean daily intakes of leucine, isoleucine and valine for adult males that were reported at 8.64, 5.01 and 5.63 g/day, respectively, once.
  Interventions: Dietary Supplement: Amino acids
- Isoleucine (Experimental): Dietary Interventions: The dose of the different BCAAs Amino acids - 5 g, is set not to exceed the mean daily intakes of leucine, isoleucine and valine for adult males that were reported at 8.64, 5.01 and 5.63 g/day, respectively, once.
  Interventions: Dietary Supplement: Amino acids
- Valine (Experimental): Dietary Interventions: The dose of the different BCAAs Amino acids- 5 g, is set not to exceed the mean daily intakes of leucine, isoleucine and valine for adult males that were reported at 8.64, 5.01 and 5.63 g/day, respectively, once.
  Interventions: Dietary Supplement: Amino acids

INTERVENTIONS:
Dietary Supplement: monosaccharides — The monosaccharides; Glucose, Fructose, Galactose and mannose, will be administrated after O.N fasting, 50gr, once.
  Arms: Fructose; Galactose; Glucose; Mannose
Dietary Supplement: Disaccharides — The Disaccharides; Lactose, Maltose and sucrose, will be administrated after O.N fasting, 50gr, once.
  Arms: Lactose; Maltose; Sucrose
Dietary Supplement: Amino acids — The Amino acids; Leucine, Isoleucine, and Valine, will be administrated after O.N fasting, 5g, once.
  Arms: Isoleucine; Leucine; Valine
Dietary Supplement: Artificial Sweeteners — The Artificial sweeteners: Saccharin, Aspartame, Sucralose and Steviol, will be administrated after O.N fasting, 300 mg, once.
  Arms: Aspartame; Saccharin; Steviol; Sucralose
Other: Control- water — Chilled water flavored with lemon juice as control
  Arms: Control

SUMMARY:
While previous atherosclerosis-related studies have focused mainly on the atherogenicity of lipids, the proposed study aims to investigate the effects of other dietary factors, i.e. monosaccharides, disaccharides, amino acids, or artificial sweeteners, on the atherogenicity of serum or macrophages. Findings from the current proposed study may shed light on yet unknown mechanisms by which the above dietary factors could affect atherosclerosis development and CVD risk and hence could possibly assist in the future development of anti-atherogenic strategies.

DETAILED DESCRIPTION:
Atherosclerosis is the underlying cause of cardiovascular diseases (CVD), the major cause of death worldwide. Atherosclerosis is an inflammatory disease of the arteries in which activated macrophages are abundant in the atherosclerotic lesions.

Macrophages play key roles during early atherogenesis. After differentiating from peripheral blood monocytes, the formed intimal macrophages take up oxidized/modified lipoproteins and are transformed into lipid-rich foam cells, the hallmark feature of early atherogenesis. In addition to lipoprotein uptake, lipid accumulation in macrophages can also result from alterations in cellular lipid metabolism, e.g. attenuated reverse lipid transport or enhanced rates of lipid biosynthesis. CVD and atherosclerosis development are significantly affected by nutritional factors. Although much progress has been made in understanding the role of different lipids (fatty acids, cholesterol, phospholipids or triglycerides) in atherosclerosis development and macrophage foam-cell formation, little is known about the potential impact of other nutrients, i.e. sugars or amino acids. For instance, hyperglycemia is known to enhance atherosclerosis development, and high glucose levels increases macrophage atherogenicity via pro-inflammatory and oxidative stress-related mechanisms. However, the role of monosaccharides other than glucose (fructose, galactose or mannose) and that of various disaccharides (maltose, sucrose or lactose) in macrophage foam-cell formation, the key event during early atherogenesis, is currently unknown. As for amino acids, a specific subgroup - the branched-chain amino acids (BCAAs), has recently been associated with increased CVD risk. The BCAA subgroup, composed of leucine, isoleucine, and valine, is characterized by an aliphatic structure of their side chains and by a common catabolic pathway. Recent reports have demonstrated an association between BCAAs, CVD and coronary artery disease (CAD). Serum BCAA levels have been positively associated with various CAD risk factors and with the development as well as the severity of CAD, even after controlling for other risk factors. Nevertheless, the role of BCAAs in atherosclerosis development and macrophage foam-cell formation is currently unclear. In recent decades, the availability and the consumption of various artificial sweeteners have increased considerably. In the USA for instance, approximately 30% of adults and 15% of children, report consumption of artificial sweeteners. Although the consumption of artificial sweeteners was previously associated with elevated risk for coronary heart disease (CHD), the effects of different artificial sweeteners, e.g. saccharin, aspartame, sucralose, steviol, cyclamate, and mannitol, on atherosclerosis development and their possible impact on macrophage foam-cell formation have not been investigated yet..

ELIGIBILITY:
Inclusion Criteria:

* Inclusion criteria will include healthy adult males between the ages of 18-50 after signing informed consent.

Exclusion Criteria:

* Exclusion criteria will include cardiovascular or pulmonary diseases, diabetes, cancer, morbid obesity (body mass index > 40 kg/m2), heavy smoking (> 20 cigarettes/day), or consumption of more than two alcoholic drinks per day.

Ages: 18 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 90 (Estimated)
Dates: Start 2016-09; Primary Completion 2018-05 (Estimated); Study Completion 2018-08 (Estimated)

PRIMARY OUTCOMES:
serum Oxidation dietary factors, i.e. monosaccharides, disaccharides, amino acids, or artificial atherogenicity of serum | 2 years
  serum oxidation level; TBARS (nmol MDA /ml)
macrophages cellular Oxidation. | 2 years
  oxidation level; TBARS (nmol MDA /mg protein)

SECONDARY OUTCOMES:
Serum lipids- Cholesterol | 2 years
  Cholesterol concentration (mg/dl)
Serum lipids- Triglycerides | 2 years
  Triglyceride concentration (mg/dl)
macrophages cellular lipids- Cholesterol | 2 years
  macrophage Cholesterol mass (mg/mg protein)
macrophages cellular lipids -Triglycerides | 2 years
  macrophage Triglyceride mass (mg/mg protein)

CONTACTS AND LOCATIONS:
Overall Officials: Tony Hayek, Prof., Principal Investigator — Rambam Health care center
Locations (1):
- Rambam Health care center, Haifa, Haifa District, Israel

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Michas G, Micha R, Zampelas A. Dietary fats and cardiovascular disease: putting together the pieces of a complicated puzzle. Atherosclerosis. 2014 Jun;234(2):320-8. doi: 10.1016/j.atherosclerosis.2014.03.013. Epub 2014 Mar 27. PMID 24727233
- [Background] Dickhout JG, Basseri S, Austin RC. Macrophage function and its impact on atherosclerotic lesion composition, progression, and stability: the good, the bad, and the ugly. Arterioscler Thromb Vasc Biol. 2008 Aug;28(8):1413-5. doi: 10.1161/ATVBAHA.108.169144. No abstract available. PMID 18650503
- [Background] Bornfeldt KE, Tabas I. Insulin resistance, hyperglycemia, and atherosclerosis. Cell Metab. 2011 Nov 2;14(5):575-85. doi: 10.1016/j.cmet.2011.07.015. PMID 22055501
- [Background] Huang Y, Zhou M, Sun H, Wang Y. Branched-chain amino acid metabolism in heart disease: an epiphenomenon or a real culprit? Cardiovasc Res. 2011 May 1;90(2):220-3. doi: 10.1093/cvr/cvr070. PMID 21502372
- [Background] Shah SH, Bain JR, Muehlbauer MJ, Stevens RD, Crosslin DR, Haynes C, Dungan J, Newby LK, Hauser ER, Ginsburg GS, Newgard CB, Kraus WE. Association of a peripheral blood metabolic profile with coronary artery disease and risk of subsequent cardiovascular events. Circ Cardiovasc Genet. 2010 Apr;3(2):207-14. doi: 10.1161/CIRCGENETICS.109.852814. Epub 2010 Feb 19. PMID 20173117
- [Background] Bhattacharya S, Granger CB, Craig D, Haynes C, Bain J, Stevens RD, Hauser ER, Newgard CB, Kraus WE, Newby LK, Shah SH. Validation of the association between a branched chain amino acid metabolite profile and extremes of coronary artery disease in patients referred for cardiac catheterization. Atherosclerosis. 2014 Jan;232(1):191-6. doi: 10.1016/j.atherosclerosis.2013.10.036. Epub 2013 Nov 12. PMID 24401236
- [Background] Yang RY, Wang SM, Sun L, Liu JM, Li HX, Sui XF, Wang M, Xiu HL, Wang S, He Q, Dong J, Chen WX. Association of branched-chain amino acids with coronary artery disease: A matched-pair case-control study. Nutr Metab Cardiovasc Dis. 2015 Oct;25(10):937-42. doi: 10.1016/j.numecd.2015.06.003. Epub 2015 Jun 14. PMID 26231617
- [Background] Yang R, Dong J, Zhao H, Li H, Guo H, Wang S, Zhang C, Wang S, Wang M, Yu S, Chen W. Association of branched-chain amino acids with carotid intima-media thickness and coronary artery disease risk factors. PLoS One. 2014 Jun 9;9(6):e99598. doi: 10.1371/journal.pone.0099598. eCollection 2014. PMID 24910999
- [Background] Swithers SE. Artificial sweeteners produce the counterintuitive effect of inducing metabolic derangements. Trends Endocrinol Metab. 2013 Sep;24(9):431-41. doi: 10.1016/j.tem.2013.05.005. Epub 2013 Jul 10. PMID 23850261
- [Background] Fung TT, Malik V, Rexrode KM, Manson JE, Willett WC, Hu FB. Sweetened beverage consumption and risk of coronary heart disease in women. Am J Clin Nutr. 2009 Apr;89(4):1037-42. doi: 10.3945/ajcn.2008.27140. Epub 2009 Feb 11. PMID 19211821
- [Result] Rom O, Aviram M. Endogenous or exogenous antioxidants vs. pro-oxidants in macrophage atherogenicity. Curr Opin Lipidol. 2016 Apr;27(2):204-6. doi: 10.1097/MOL.0000000000000287. No abstract available. PMID 26959710